CLINICAL TRIAL: NCT05219175
Title: MDMA-Assisted Therapy 6 to 12 Months After Childbirth for People With Co-occurring Opioid Use and Post Traumatic Stress Disorders
Brief Title: MDMA for Co-occurring PTSD and OUD After Childbirth
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Multidisciplinary Association for Psychedelic Studies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUSOU1
Record Dates: First submitted 2022-01-02; First posted 2022-02-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Stress Disorders, Post-Traumatic; Opioid Use Disorder
Keywords: PTSD; Opioid Use Disorder; Addiction; MDMA; Psychedelic Assisted Therapy; Maternal Infant Bonding
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Opioid-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Intervention Model Description: Open label study comparing outcomes before and after treatment with MDMA Assisted Therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Co-occurring PTSD and OUD prior and after treatment with MDMA Assisted Therapy (Experimental): The intervention is MDMA Assisted Therapy focused on PTSD and three experiment sessions with the first session using an initial dose of 100 mg MDMA HCL (~80 mg MDMA) with supplemental dose of 40 mg MDMA HCL (~35 mg MDMA). Total dose range for the first session is 100 mg MDMA HCL (~80 mg MDMA) to 140 mg MDMA HCL (~115 mg MDMA).The second and third sessions may use an initial dose of 120 mg MDMA HCL (~100 mg MDMA) with a supplemental dose of 60 mg MDMA HCL (~50 mg MDMA) for a total dose range of 120 mg MDMA HCL (~100 mg MDMA) to 180 mg MDMA HCL (~160 mg MDMA)
  Total cumulative dose range for the three sessions is 340mg MDMA HCL (~280 mg MDMA) to 500 mg MDMA HCL (~435 mg MDMA)
  Interventions: Drug: MDMA Assisted Therapy

INTERVENTIONS:
Drug: MDMA Assisted Therapy — The intervention is MDMA Assisted Therapy focused on PTSD and three experiment sessions with the first session using an initial dose of 100 mg MDMA HCL (~80 mg MDMA) with supplemental dose of 40 mg MDMA HCL (~35 mg MDMA). Total dose range for the first session is 100 mg MDMA HCL (~80 mg MDMA) to 140 mg MDMA HCL (~115 mg MDMA).The second and third sessions may use an initial dose of 120 mg MDMA HCL (~100 mg MDMA) with a supplemental dose of 60 mg MDMA HCL (~50 mg MDMA) for a total dose range of 120 mg MDMA HCL (~100 mg MDMA) to 180 mg MDMA HCL (~160 mg MDMA)
  Total cumulative dose range for the three sessions is 340mg MDMA HCL (~280 mg MDMA) to 500 mg MDMA HCL (~435 mg MDMA)

SUMMARY:
This is an open-label study of the use of MDMA Assisted Therapy for postpartum people with co-occurring Post Traumatic Stress Disorder (PTSD) and Opioid Use Disorder (OUD). The study protocol has been adapted from the Phase 3 studies sponsored by the Multidisciplinary Association for Psychedelic Studies (MAPS) for PTSD. Due to the high rate of concurrence of PTSD and OUD, people with OUD may experience great benefit from the treatment of their PTSD with MDMA-assisted therapy based on the phase 2 and 3 studies for PTSD. Use of MDMA-assisted therapy in this population has the potential to be of benefit for their OUD and maternal- infant attachment.

This study will serve to explore the feasibility and safety of offering MDMA-assisted therapy for treatment of PTSD in postpartum people with opioid use disorder. The CAPs 5 (PTSD) is the primary outcome, the Timeline Follow-Back (TLFB) for opioid use is the secondary outcome and other assessments of opioid use disorder, effects on maternal-infant attachment, social connectedness and other mental health outcomes are exploratory. The study will be conducted at the University of New Mexico Health Sciences Center located in Albuquerque New Mexico. In addition to northern New Mexico being an epicenter of the current opioid use disorder epidemic in the United States there is a long-standing history of multigenerational use of illicit opioids in many communities of northern New Mexico. There are high rates of opioid use disorder on pregnancy and accompanying Neonatal Opioid Use Withdrawal Syndrome (NOWS) in Albuquerque, Santa Fe, and surrounding communities.

DETAILED DESCRIPTION:
Protocol Synopsis MDMA-Assisted Therapy 6 to 12 months After Childbirth for People with Co-occurring Opioid Use and Post Traumatic Stress Disorders

Protocol IUSOU1:

Rationale Introduction

Background and Previous Research Data

Opioid use disorder

Opioid use disorder has reached epidemic levels in the United States and is now common in pregnant and postpartum people From 1999 to 2014 the delivery-related hospital admissions of people with opioid use disorder more than quadrupled from 1.5 to 6.5 per 1,000 delivery hospitalizations. New Mexico is one of the epicenters of the opioid use epidemic. 12.8 newborns per 1000 births in New Mexico were diagnosed with Neonatal Opioid Withdrawal Syndrome in 2018. The standard of care for Opioid Use Disorder (OUD) is the use of medication for opioid use disorder (MOUD) that was either initiated during the pregnancy or was already being taken at the time of conception. MOUD is effective at improving maternal and neonatal outcomes, however postpartum relapse is common and carries an increased risk of fatal overdose. By having the use of MOUD as an inclusion criteria we are selecting for a group of people that has a greater chance of being stable throughout the study period and at lower risk for opioid overdose than individuals who relapse and are not on MOUD.

Post-Traumatic Stress Disorder

Psychological trauma is a common antecedent of addiction, and a trauma-informed approach is integral to substance misuse care. The high rates of childhood sexual abuse and rape are factors resulting in high rates of Post Traumatic Stress Disorder (PTSD) among pregnant and postpartum people. PTSD occurs in some individuals that are exposed to an event that is perceived to result in serious injury, sexual violence or an actual or possible threat to life. Intrusive symptoms such as nightmares, flashbacks, emotional distress or physical reactivity can then recur when the traumatic event is persistently re-experienced leading to avoidance of trauma-related thoughts, feelings or reminders of the events which act as "triggers" of symptoms. The individual's life is adversely affected by negative alterations in mood and thought including the somatic symptoms of increased arousal and reactivity (e.g. hypervigilance, heightened startle reaction, and difficulty sleeping). PTSD is a serious disorder that commonly has a negative impact on an individual's quality of life including impairing their ability to work and maintain relationships and it is associated with increased substance use, depression and suicide. Symptoms must persist for at least a month at sufficient intensity to be diagnosed as PTSD, however they are often severe, last for many years and can be resistant to treatment.

PTSD can be treated with behavioral or medication therapies, however the treatments for PTSD are often not included in the services offered by perinatal substance use programs. The 2020 Guidelines from International Society for Traumatic Stress Studies include strong recommendations for the use of cognitive processing therapy, cognitive therapy, EMDR (Eye Movement Desensitization and Reprocessing), prolonged exposure and cognitive behavioral therapy with a trauma focus for adults with PTSD. Selective Serotonin Reuptake Inhibitors (SSRIs) have a modest effect on symptom reduction however they are often used long term without achieving a resolution of PTSD.

MDMA

MDMA (3, 4-Methylenedioxymethamphetamine) has received breakthrough drug status from the FDA for the treatment of PTSD. MDMA is a monoamine releaser and re-uptake inhibitor with indirect effects on neurohormone release. MDMA has a more complex neurochemical mechanism than classical psychedelics involving increased release of serotonin, dopamine, noradrenaline and oxytocin. Activation of the 5-hydroxytryptamine receptor 1A (5-HT1a) and 5-hydroxytryptamine receptor 1B (5-HT1b) receptors decreases feeling of anxiety and depression and reduces amygdala mediated fear response. These effects are accompanied by increased empathy, emotional closeness and compassion. Effects on the alpha-2 receptor are potentially beneficial in psychotherapy by reducing trauma associated hypervigilance mitigated by norepinephrine. The release of oxytocin, the hormone promoting maternal infant bonding, is hypothesized to increase empathy, feelings of "closeness; and decrease the fear activity activated in the amygdala.15,16 The neurocognitive effects of MDMA- assisted therapy have been proposed to be mediated via memory reconsolidation and fear extinction by reducing activation in the insula and amygdala which are involved with the expression and fear and anxiety. A functional Magnetic Resonance Imaging MRI study of subjects administered MDMA demonstrated a decrease in insula network connectivity lending support to the hypothesis that this is a mechanism for the effects of MDMA.

The combined neurobiological effects of MDMA reduce defenses and fear of emotional injury, enhance communication and introspection. And can increase empathy and compassion allowing for a psychological state that enhances successful trauma processing during psychotherapy.. MDMA has demonstrated benefit for treatment resistant PTSD in a series of phase 2 studies of MDMA-assisted therapy sponsored by the Multidisciplinary Association for Psychedelic Studies. In pooled analysis of six phase 2 randomized controlled trials of MDMA-assisted therapy for long term PTSD, more participants in the active group (54.2%) did not meet DSM-IV (Diagnostic Manual of Mental Disorders) PTSD diagnostic criteria than the control group (22.6%) after two MDMA sessions. Based on historical comparison MDMA appears to be more effective than the two FDA approved Selective Serotonin Reuptake Inhibitor (SSRI) medications (sertraline and paroxetine) . The processing of trauma during MDMA-assisted therapy may produce additional lasting changes by increasing the individual's personality trait of openness.

MDMA may be of benefit to people for opioid use disorder secondary to resolving or improving PTSD symptoms or by a pathway independent of PTSD. Although published research regarding the use of MDMA for substance use disorders is limited to a single small study involving alcohol use disorder described below20 there is a growing literature involving the use of classic psychedelics (e.g. psilocybin and LSD). Psilocybin has shown promise in the treatment of tobacco and alcohol use disorders and is being studied for opioid and cocaine use disorders. A novel psychedelic ibogaine has been reported as a specific treatment for opioid use disorder, however there have not been any randomized controlled trials. Lysergic Acid Diethylamide (LSD) was extensively studied as a treatment for alcohol use disorder in the 1960s and 1970s. A meta-analysis of six randomized controlled trials including 536 subjects demonstrated a beneficial effect of LSD on alcohol misuse (OR, 1.96; 95% Confidence Interval (CI), 1.36-2.84; p = 0.0003). Although rigorous prospective trials are lacking, the use of plant derived psychedelics for substance use disorders additionally includes peyote in the Native American church for alcohol use disorder in the United States and Ayahuasca for cocaine and other substance use disorders in Peru and Brazil.

The classic psychedelics work primarily at the level of the 5-HT2A receptor where they decrease activity in the brain's default mode network which is correlated with "ego dissolution". Although classic psychedelics are showing benefit for addiction there are postpartum people with opioid use disorder who may not desire the experiences of "ego dissolution" and mystical experience during the postpartum period. MDMA has psychedelic effects however it does not usually lead to the profound states of ego dissolution and "mystical experiences" that are associated with the positive effects of the classic psychedelics and detected by the Mystical Experience Questionnaire (MEQ-30). The first study of MDMA for a substance use disorder is the Bristol Imperial MDMA in Alcoholism Study (BIMA) which demonstrated the feasibility of MDMA treatment after community based alcohol detoxification. A follow-up study of alcohol consumption after MDMA treatment for PTSD demonstrated that alcohol consumption since study enrollment decreased among 22 participants (40.0%), stayed the same for 17 participants (30.9%), and increased for 2 participants (3.6%) compared to prior to study enrollment.

OUD, PTSD, and MDMA

OUD and PTSD are strongly associated comorbid disorders. The association between these conditions may be due to traumatic life events leading to PTSD which are "self-medicated" with the opioid, however the lifestyle of individuals with opioid use disorder may also predispose to an increased likelihood of traumatic events. In pregnant woman with high rates of adverse childhood events, it is these traumatic events that usually precede the development of OUD. However, trauma that occurs after they have OUD may intensify their PTSD symptoms. An Australian study of individuals with heroin dependence demonstrated that 90% had serious trauma in the life history and 40% had PTSD. The U.S. National Comorbidity Survey of the general population estimated a lifetime prevalence rate of PTSD of 6.8% and current past year PTSD prevalence of 3.5%.The lifetime prevalence of PTSD among men was 3.6% and among women was 9.7%. Woman have higher 12 month prevalence rates of PTSD of 5.2% compared to 1.8% among men.

Racial trauma may contribute to PTSD either due to a major life event occurring directly due to racism including hate crimes or workplace harassment or due to a series of subtler lifelong occurrences that are the result of micro aggressions and implicit racial bias. To identify these sources of trauma newer assessment instruments have been developed including the UConn Racial/Ethnic Stress and Trauma Survey and a short version which has been used by MDMA therapists. A culturally informed approach to MDMA assisted therapy for PTSD includes cultural diversity on the treatment team, outreach to communities of color, and development of a setting including music and artwork that is culturally sensitive and appropriate. This can include conveying an appreciation that most psychedelic therapies have their roots in the plant medicine of indigenous healers (e.g. psilocybin, peyote and ayahuasca) and that the approach to using synthesized psychedelics that are not plant derived (e.g. MDMA and ketamine) can still integrate learning from these indigenous practices.

Maternal PTSD and substance use disorders have been proposed as mechanisms of intergenerational trauma transmission through their effect on maternal infant bonding. The disruption of maternal attachment leads to an increased risk of the child developing substance use disorder. Treating maternal PTSD during pregnancy or postpartum has the theoretical potential to decrease the likelihood of the infant developing a substance use disorder during adolescence or adulthood. As MDMA appears to be effective in the treatment of PTSD in other populations, a feasibility study of the use of MDMA-assisted therapy in postpartum people with OUD has great potential to benefit the infant as well as the mother. Use of MDMA during pregnancy or during breastfeeding presents an unacceptable level of maternal and neonatal risk due to the lack of safety data, however studies of postpartum people at the University of New Mexico have demonstrated that the average time for stopping breastfeeding in this group was three weeks postpartum therefore offering MDMA- assisted therapy for PTSD at 6-12 months of age would only exclude a small proportion of people due to ongoing breastfeeding.

Although the likelihood of benefit for opioid use disorder from MDMA experimental sessions may not be associated with higher scores on the MEQ-30, there are other instruments that can assess the effect of the experience on the participant. The Challenging Experience Questionnaire has been used to assess the effects of challenging emotions such as fear or paranoia which may be a negative predictor of a positive response from the sessions.The CEQ does not address the issue of how the challenging experience was resolved. Challenging experiences may potentially facilitate transformation through a "pivotal state" that may increase neuroplasticity and deep learning. Stanislav Grof, a founder of transpersonal psychology and author of "LSD Psychotherapy" felt that challenging psychedelic experiences were of benefit in supporting psychological transformation.The recently developed Emotional Breakthrough Inventory (EBI) was developed to complement the MEQ-30 and CEQ and to look at the participant's ability to achieve a breakthrough experience by overcoming challenging emotions and memories.Understanding the psychological processes that support positive change such as resolution of PTSD or maintenance of remission for opioid use disorder is an exploratory objective.

Indications being studied:

Co-occurring Post Traumatic Stress Disorder and Opioid User Disorder

Treatment Proposal and Rationale

Due to the high rate of concurrence of PTSD and OUD these people may experience great benefit from the treatment of their PTSD with MDMA-assisted therapy based on the phase 2 and 3 studies for PTSD. Use of MDMA-assisted therapy in this population has the potential to be of benefit for their OUD and maternal- infant attachment. This open-label study will serve to explore the feasibility and safety of offering MDMA-assisted therapy for treatment of PTSD in postpartum people with opioid use disorder. The CAPs 5 (PTSD) is the primary outcome, the Timeline Follow-Back (TLFB) for opioid use is the secondary outcome and other assessments of opioid use disorder, effects on maternal-infant attachment, social connectedness and other mental health outcomes are exploratory.

Study Design This is a single site open-label feasibility study to assess the safety and effectiveness of MDMA-assisted therapy in 15 people who are between six to twelve months after childbirth with co-existing opioid use disorder (OUD) and postt-raumatic stress disorder (PTSD). The therapy teams will have received training in MDMA-assisted therapy provided by the Multidisciplinary Association for Psychedelic Studies (MAPS).

For the first medication sessions participants will receive a dose of 100 mg MDMA Hydrochloric acid (HCL) (~80 mg MDMA ), followed by a supplemental 40 mg MDMA HCL (~35 mg MDMA) dose two hours after receiving the initial dose unless tolerability issues emerge with the first dose or the participant declines. MDMA is administered during the Treatment Period with manualized therapy in three open-label monthly Experimental Sessions. This ~12-week Treatment Period is preceded by two three Preparatory Sessions. During the Treatment Period, each Experimental Session is followed by three Integrative Sessions of non-drug therapy. The second and third medication sessions may use 120 mg MDMA Hydrochloric acid (HCL) (~100 mg MDMA ),followed by a supplemental 60 mg MDMA HCL (~50 mg MDMA) dose two hours after receiving the initial dose unless tolerability issues emerge with the first dose or the participant declines.

For each participant, the study will consist of:

* Screening Period: phone screen, informed consent, eligibility assessment, and enrollment if eligible
* Preparatory Period with Enrollment Confirmation: medication tapering, Preparatory Sessions and Baseline assessments
* Treatment Period: three monthly Medication Sessions and associated Integrative Sessions over ~12 weeks
* Follow-up Period and Study Conclusion:

The 1-month Primary Outcome visit will occur 4 weeks (+/- 2 weeks) after the last study session.

• At 6 months after the last study session a final assessment will occur for the PTSD and OUD outcomes.

Psychotherapeutic Model for MDMA Assisted therapy for PTSD and OUD

The manual for MDMA-assisted therapy of PTSD uses a nondirective approach with a focus on using empathetic presence and listening. The approach is person centered therapy where the participant uses their own inner healing intelligence to guide their therapy. In this study the participants have opioid use disorder which has been stable on MOUD (buprenorphine or methadone) for at least three months. The study will use motivational interviewing (MI) techniques, to guide the initiation of the therapy for opioid use disorder. MI is also a patient centered approach rooted in empathic listening and can address the common issue of ambivalence of entering a trauma centered therapy. Therapists may choose approaches that use the tools of acceptance and commitment therapy (ACT) , motivational enhancement therapy, and mindfulness among other approaches that have been used with psychedelic assisted therapies. The investigators are following the approach of MDMA-assisted therapy manual for PTSD, which allows for elements of other therapeutic approaches to be applied as long as they are done so within the guidelines of the Manual. The study will not attempt to manualize the additional elements of opioid use disorder therapy. The investigators will maintain a record of the psychotherapeutic context of the preparatory and integration sessions.

Recruitment and Participant Population Subject Recruitment People using buprenorphine will primarily be recruited during pregnancy from the Milagro Perinatal Substance Use Program at the University of New Mexico (UNM) and the GRACE Program at Lovelace Women's Hospital in Albuquerque New Mexico. These two programs care for almost all the pregnant people using buprenorphine or methadone for MOUD during pregnancy in the greater Albuquerque area. The Milagro program cares for approximately 150 pregnant people per year of which about 90% (n=120) have opioid use disorder on MOUD and about 60% are using methadone (n=72) and 40% buprenorphine (n=48). The people in the Milagro program are about 90% Hispanic, 10% non-Hispanic White with an occasional Native American woman. The Grace program cares for about 25 pregnant people a year who are using buprenorphine. A third recruitment site in Albuquerque will be the University of New Mexico (UNM) FOCUS program which collaborates with Milagro by providing well-child and developmental care to infants born to the people in Milagro, as well as other people with substance use disorders, and offers ongoing buprenorphine to people after childbirth. The PI for this study, Larry Leeman MD, is the Medical Director for Milagro. . Participation in the study will also be offered to pregnant and postpartum people prescribed buprenorphine who receive care in Santa Fe, sixty miles north of Albuquerque. Information regarding the study will be provided to physicians offering prenatal care in Santa Fe, however screening and all study procedures will occur at UNM. The research team will carefully assess the potential participant's willingness and motivation to make the sixty-mile drive to Albuquerque and back for all required in-person study visits prior to enrollment in the study.

Statistical Analysis The primary outcome is the change from baseline in the Total Severity Score from the CAPS 5 until 1 month after the 3rd medication visit. The investigators will perform paired T tests for the two assessment periods to see if the confidence interval overlaps between the two groups. The investigators will also compare the effect size as measured by CAPS 5 in this cohort with OUD compared to the MAPP1 and MAPP2 cohorts which had OUD as an exclusion criteria.

The secondary outcome is to evaluate the effect of MDMA-assisted therapy for PTSD on the Opioid Use by the TLFB assessment of the number of days of illicit opioid use in the baseline thirty-day period compared to the thirty-day period preceding the 6-month follow-up visit. As a normal a distribution curve is not anticipated , the nonparametric Wilcoxon signed rank test will be used.

For the exploratory outcomes the investigators will collect estimates of Hedges g effect size for continuous measures, to determine the sample size of a powered study for any of the measures studied.

An exploratory objective is to evaluate the effect of MDMA assisted therapy on maternal-infant-bonding, attachment and parenting as measured by multiple questionnaires assessments and use of the Still Face Paradigm (SFP), a well-known, objective measure of bonding and attachment, to obtain video assessment of the mother as she is interacting with her baby. The SFP videos are recorded prior to study initiation, on the morning after each MDMA session and after completion of the study. Participants may decide not to participate in the SFP video assessments without affecting their participation in the primary study of MDMA-AT for OUD and PTSD .

A qualitative analysis will be included based on a structured interview that will occur with all participants between 4-8 weeks after the 3rd experimental session. The investigators will work with a UNM social scientist which may be a PhD Psychologist who has previously collaborated with this team in prior PTSD in pregnancy research.

ELIGIBILITY:
Inclusion Criteria:

* Potential participants are eligible to enroll in the protocol if they:

  1. Are at least 18 years old.
  2. Have opioid use disorder and are using daily oral methadone of 180 mg or less, or sublingual buprenorphine (or buprenorphine with naloxone in 4:1 ratio) of 24 mg or less. Assessed as stable for at least 3 months based upon review of the University of New Mexico Milagro and FOCUS program medical records or direct communication with the participant's buprenorphine or methadone prescriber.
  3. Are fluent in speaking and reading English. This criteria is needed as the protocol requires two therapists that have specific training and it would be very difficult to identify two therapists fluent in another language
  4. Are able to swallow pills.
  5. Agree to have study visits recorded, including Experimental Sessions, Independent Rater assessments by an on-site Independent Rater for CAPS-5, and non-drug therapy sessions.
  6. Must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
  7. Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
  8. If able to become pregnant, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session. Adequate birth control methods include intrauterine device (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e., condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom). Not able to become pregnant is defined as permanent sterilization or postmenopausal.
  9. Agree to the lifestyle modifications described in Section 3.0 above:

     Medical History
  10. At Screening, meet DSM-5 criteria for current moderate to severe PTSD with a symptom duration of 6 months or longer.
  11. At Screening, meet DSM-5 criteria for Opioid Use Disorder.
  12. At Screening, have had PTSD symptoms for at least three months and at least moderate PTSD symptoms in the last month based on PCL-5 total score of 40 or greater.
  13. May have well-controlled hypertension that has been successfully treated with anti-hypertensive medicines, if they pass additional screening to rule out underlying cardiovascular disease
  14. May have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
  15. At Baseline, have at least moderate PTSD per CAPS-5 and symptoms in the last month constituting a CAPS-5 Total Severity Score of 28 or greater
  16. May have current mild alcohol or cannabis use disorder (meets 2 or 3 of 11 diagnostic criteria per DSM-5) or moderate alcohol or cannabis use disorder in early remission for the 3 months prior to enrollment (meets 5 of 11 diagnostic criteria per DSM-5).
  17. May have a history of or current Diabetes Mellitus (Type 2) if additional screening measures rule out underlying cardiovascular disease, if the condition is judged to be stable on effective management, and with approval by the study physician.
  18. May have hypothyroidism if taking adequate and stable thyroid replacement medication.
  19. May have a history of, or current, glaucoma if approval for study participation is received from an ophthalmologist.

Exclusion Criteria (partial):

* Potential participants are ineligible to enroll in the protocol if they:

  1. Are not able to give adequate informed consent.
  2. Prisoners will be excluded
  3. Are likely, in the investigator's opinion and via observation during the Preparatory Period, to be re-exposed to their index trauma, lack social support, or lack a stable living situation.
  4. Have any current problem which, in the opinion of the investigator or study physician, might interfere with participation.
  5. A 12 Lead EKG demonstrates QTc greater than 460 msec at time of screening for any potential participant or for the participants using methadone on an EKG obtained within 72 hours of each MDMA treatment session. An abnormal EKG may be repeated once to confirm the presence of QTc prolongation. 460 msec used as the upper acceptable limit as this study only includes women and the level of QTc that is considered abnormal is 10-20 msec longer for women.

     Psychiatric History

  7. Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment. 8. Have a history of or a current primary psychotic disorder, bipolar disorder 1 assessed via MINI and clinical interview or dissociative identity disorder assessed via structured clinical interview (SCID).

  9. Have a current eating disorder with active purging assessed via MINI and clinical interview.

  10. Have current major depressive disorder with psychotic features assessed via MINI.

  11. Have a current moderate (not in early remission in the 3 months prior to enrollment based on meeting 4 or 5 of 11 diagnostic criteria per DSM-5) or severe alcohol or cannabis use disorder within the 6 months prior to enrollment (meets at least 6 of 11 diagnostic criteria per DSM-5).

  12. Have an active illicit (other than cannabis or opioids) or prescription drug substance use disorder at any severity within 3 months prior to enrollment.

  13. If there has been a diagnosis of moderate or severe cannabis use disorder within the last six months prior to enrollment, then the participant will need to have tapered off cannabis prior to the time of enrollment in the study and have either entered abstinence, limited cannabis use, or mild cannabis disorder. Mild cannabis use disorder or cannabis use alone are not exclusion criteria, however there can be no use in the 24 hours prior to the medication session.

  14. Have current Personality Disorders Cluster A (paranoid, schizoid, schizotypal),) assessed via SCID-5-PD 15. Investigators will exclude potential participants with high risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation (e.g., evidence of serious personality disorder, antisocial behavior, serious current stressors, or lack of meaningful social support) 16. Any participant presenting current serious suicide risk, as determined through psychiatric interview, responses to C-SSRS, and clinical judgment of the investigator will be excluded; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior, in the judgment of the investigator, will not be enrolled.

Medical History

17. Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate.

19. Have uncontrolled essential hypertension using the standard criteria of the American Heart Association (values of 140/90 milligrams of Mercury [mmHg] or higher assessed on three separate occasions).

20. Have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease.

21. Have a history of arrhythmia, other than occasional premature atrial contractions (PACs) or PVCs in the absence of ischemic heart disease, within 12 months of screening.

23. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).

24. Require use of concomitant medications that prolong the QT/QTc interval during Experimental Sessions. Refer to Protocol Section _12___: Concomitant Medications.

25. Have symptomatic liver disease or have significant liver enzyme elevations. 26. Have history of hyponatremia or hyperthermia. 27. Weigh less than 48 kilograms (kg). 29. Are pregnant or are able to become pregnant and are not practicing an effective means of birth control.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
PTSD | 4 weeks after 3rd experimental session
  CAPS-5

SECONDARY OUTCOMES:
Opioid Use Disorder | 6 months after 3rd Experimental Sessions
  TLFB ( Timeline Followback)

OTHER OUTCOMES:
Effect on nonopioid substance use disorders | 1-6 months after 3rd Experimental Session
  TLFB

CONTACTS AND LOCATIONS:
Overall Officials: Hadya Khawaja, MS, CIP, Study Director — UNM Health Sciences Human Research Protections Program
Locations (1):
- University of New Mexico Health Sciences, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mitchell JM, Bogenschutz M, Lilienstein A, Harrison C, Kleiman S, Parker-Guilbert K, Ot'alora G M, Garas W, Paleos C, Gorman I, Nicholas C, Mithoefer M, Carlin S, Poulter B, Mithoefer A, Quevedo S, Wells G, Klaire SS, van der Kolk B, Tzarfaty K, Amiaz R, Worthy R, Shannon S, Woolley JD, Marta C, Gelfand Y, Hapke E, Amar S, Wallach Y, Brown R, Hamilton S, Wang JB, Coker A, Matthews R, de Boer A, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted therapy for severe PTSD: a randomized, double-blind, placebo-controlled phase 3 study. Nat Med. 2021 Jun;27(6):1025-1033. doi: 10.1038/s41591-021-01336-3. Epub 2021 May 10. PMID 33972795
- [Result] Haight SC, Ko JY, Tong VT, Bohm MK, Callaghan WM. Opioid Use Disorder Documented at Delivery Hospitalization - United States, 1999-2014. MMWR Morb Mortal Wkly Rep. 2018 Aug 10;67(31):845-849. doi: 10.15585/mmwr.mm6731a1. PMID 30091969
- [Result] Nardou R, Lewis EM, Rothhaas R, Xu R, Yang A, Boyden E, Dolen G. Oxytocin-dependent reopening of a social reward learning critical period with MDMA. Nature. 2019 May;569(7754):116-120. doi: 10.1038/s41586-019-1075-9. Epub 2019 Apr 3. PMID 30944474
- [Result] Mithoefer MC, Feduccia AA, Jerome L, Mithoefer A, Wagner M, Walsh Z, Hamilton S, Yazar-Klosinski B, Emerson A, Doblin R. MDMA-assisted psychotherapy for treatment of PTSD: study design and rationale for phase 3 trials based on pooled analysis of six phase 2 randomized controlled trials. Psychopharmacology (Berl). 2019 Sep;236(9):2735-2745. doi: 10.1007/s00213-019-05249-5. Epub 2019 May 7. PMID 31065731
- [Result] Sessa B, Higbed L, O'Brien S, Durant C, Sakal C, Titheradge D, Williams TM, Rose-Morris A, Brew-Girard E, Burrows S, Wiseman C, Wilson S, Rickard J, Nutt DJ. First study of safety and tolerability of 3,4-methylenedioxymethamphetamine-assisted psychotherapy in patients with alcohol use disorder. J Psychopharmacol. 2021 Apr;35(4):375-383. doi: 10.1177/0269881121991792. Epub 2021 Feb 18. PMID 33601929
- [Result] Bogenschutz MP, Johnson MW. Classic hallucinogens in the treatment of addictions. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Jan 4;64:250-8. doi: 10.1016/j.pnpbp.2015.03.002. Epub 2015 Mar 14. PMID 25784600
- [Result] Reiff CM, Richman EE, Nemeroff CB, Carpenter LL, Widge AS, Rodriguez CI, Kalin NH, McDonald WM; the Work Group on Biomarkers and Novel Treatments, a Division of the American Psychiatric Association Council of Research. Psychedelics and Psychedelic-Assisted Psychotherapy. Am J Psychiatry. 2020 May 1;177(5):391-410. doi: 10.1176/appi.ajp.2019.19010035. Epub 2020 Feb 26. PMID 32098487
- [Result] Winkelman M. Psychedelics as medicines for substance abuse rehabilitation: evaluating treatments with LSD, Peyote, Ibogaine and Ayahuasca. Curr Drug Abuse Rev. 2014;7(2):101-16. doi: 10.2174/1874473708666150107120011. PMID 25563446
- [Result] Meulewaeter F, De Pauw SSW, Vanderplasschen W. Mothering, Substance Use Disorders and Intergenerational Trauma Transmission: An Attachment-Based Perspective. Front Psychiatry. 2019 Oct 18;10:728. doi: 10.3389/fpsyt.2019.00728. eCollection 2019. PMID 31681040
- [Result] Danovitch I. Post-traumatic stress disorder and opioid use disorder: A narrative review of conceptual models. J Addict Dis. 2016 Jul-Sep;35(3):169-79. doi: 10.1080/10550887.2016.1168212. Epub 2016 Mar 24. PMID 27010975
- [Result] Mills KL, Lynskey M, Teesson M, Ross J, Darke S. Post-traumatic stress disorder among people with heroin dependence in the Australian treatment outcome study (ATOS): prevalence and correlates. Drug Alcohol Depend. 2005 Mar 7;77(3):243-9. doi: 10.1016/j.drugalcdep.2004.08.016. PMID 15734224